CLINICAL TRIAL: NCT02697799
Title: A Randomized Trial of Recruitment Strategies for Research Participation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Massachusetts General Hospital (Other); Washington University School of Medicine (Other); M.D. Anderson Cancer Center (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Scott Halpern, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 823491
Record Dates: First submitted 2016-02-25; First posted 2016-03-03 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Incentives; Research Ethics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-level recruitment strategy (Experimental): Subjects in this group will receive pre-consent messaging and a consent form with a high-level recruitment strategy for research participation in the parent study. The consent form will provide information on the first page, under the header that describes the purpose of the study, as well as in the consent sections describing the cost to participate in the study.
  Interventions: Behavioral: High-level recruitment strategy consent form
- Mid-level recruitment strategy (Experimental): Subjects in this group will receive pre-consent messaging and a consent form with a mid-level recruitment strategy for research participation in the parent study. The consent form will provide information on the first page, under the header that describes the purpose of the study, as well as in the consent sections describing the cost to participate in the study.
  Interventions: Behavioral: Mid-level recruitment strategy consent form
- No modified recruitment strategy (No Intervention): Subjects in this group will receive consent form without a modified recruitment strategy for research participation in the parent study.

INTERVENTIONS:
Behavioral: High-level recruitment strategy consent form — Patients will be exposed to pre-consent messaging and a consent form that includes supplemental information describing a high-level recruitment strategy
  Arms: High-level recruitment strategy
Behavioral: Mid-level recruitment strategy consent form — Patients will be exposed to pre-consent messaging and a consent form that includes supplemental information describing a mid-level recruitment strategy
  Arms: Mid-level recruitment strategy

SUMMARY:
In a multicenter, randomized clinical trial of attitudes towards research participation, we will evaluate the ethics, effectiveness, and cost- effectiveness of three recruitment strategies for research participation in a mobility trial among hospitalized patients and a smoking cessation trial among patients with depression.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for parent RCT
2. 18 years or older
3. No prior knowledge of recruitment strategies used for this trial
4. Speaks English

Exclusion Criteria:

1)Prior knowledge of recruitment strategies used for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1296 (Actual)
Dates: Start 2016-08; Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the proportion of people assigned to each recruitment strategy that consent to participate in the two parent RCTs. | Immediate- Several Days
  Consent rates in each of the two parent RCTs

SECONDARY OUTCOMES:
Attitudes towards research | Immediate
  Attitudes towards research will be measured using the Research Attitudes Questionnaire-7 (RAQ-7). Originally designed with 11 items, a shorter 7-item version (RAQ-7) has been shown to have improved internal consistency and factorial validity.
Attention to informed consent | Immediate
  We will assess the amount of time patients spend reading each part of the parent RCT consent forms. On-site research coordinators will facilitate the collection of this data as patients read the document via the recruitment strategy study's electronic database.
Perceived risks of the research | Immediate
  Perceived risks of the research will be measured by the 9-item compared riskiness scale, which assesses perceptions of research risk. Using this approach, patients compare their assessment of the riskiness of the RCTs to other salient and more commonly encountered risks. Such comparative assessments have been shown to be less susceptible to errors in scale calibration than isolated ratings of risks.
Incidence of therapeutic misconceptions | Immediate
  We will assess patients' ability to distinguish research from individualized patient care by measuring rates of therapeutic misconception across recruitment strategies among patients considering participation in the parent RCTs. We will assess this outcome with a 4-item tool developed by Dr. Scott Kim, which has been used for similar purposes in several research contexts.
Understanding of the trial | Immediate
  To assess whether increased attention translates into improved understanding of the parent RCTs, we will use a 6-item Trial Elements Quiz, featuring core elements of the parent RCTs' consent form.
Perceptions of influence or coercion | Immediate
  To measure general perception of coercion and voluntariness of research participation, we will use the five-item Perceived Coercion Scale of the MacArthur Admission Experience Survey. The true/false scale is tailored to measure patients' perceptions of coercion in the inpatient psychiatric treatment admission process; we have edited the wording to make it relevant to participation in the parent RCTs.
Retention through the end of treatment sessions | 8 - 27 weeks
  We will assess the impact of the recruitment strategies on retention status in the protocol of the parent RCTs.

CONTACTS AND LOCATIONS:
Overall Officials: Scott D Halpern, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krutsinger DC, McMahon J, Stephens-Shields AJ, Bayes B, Brooks S, Hitsman BL, Lubitz SF, Reyes C, Schnoll RA, Ryan Greysen S, Mercede A, Patel MS, Reale C, Barg F, Karlawish J, Polsky D, Volpp KG, Halpern SD. Randomized evaluation of trial acceptability by INcentive (RETAIN): Study protocol for two embedded randomized controlled trials. Contemp Clin Trials. 2019 Jan;76:1-8. doi: 10.1016/j.cct.2018.11.007. Epub 2018 Nov 8. PMID 30414865
- [Result] Halpern SD, Chowdhury M, Bayes B, Cooney E, Hitsman BL, Schnoll RA, Lubitz SF, Reyes C, Patel MS, Greysen SR, Mercede A, Reale C, Barg FK, Volpp KG, Karlawish J, Stephens-Shields AJ. Effectiveness and Ethics of Incentives for Research Participation: 2 Randomized Clinical Trials. JAMA Intern Med. 2021 Nov 1;181(11):1479-1488. doi: 10.1001/jamainternmed.2021.5450. PMID 34542553

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT02697799/Prot_SAP_000.pdf